CLINICAL TRIAL: NCT00914472
Title: A Randomized Non-inferiority Clinical Trial of Heparin Produced by Hipolabor Laboratory(PARINEX®) in Comparation With Heparin Produced by APP PHARMACEUTICALS in Patients With Chronic Renal Failure.
Brief Title: Comparison of Two Heparin Formulations in Patients With Chronic Renal Failure.
Acronym: HEPHIP0509
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica Pesquisa e Desenvolvimento Ltda
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HEPHIP0509; Version 01
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2009-12

CONDITIONS: Thrombus
Keywords: Preventing the thrombi formation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Heparin - Hipolabor
  Interventions: Biological: Heparin sodium - Hipolabor
- Ative comparator (Active Comparator): Heparin - APP
  Interventions: Biological: heparin sodium - APP

INTERVENTIONS:
Biological: heparin sodium - APP — Heparin 5000 IU / mL
  Arms: Ative comparator
Biological: Heparin sodium - Hipolabor — Heparin 5000 IU / mL
  Arms: Test

SUMMARY:
Investigate, through a randomized, open, parallel and comparative, non-inferiority of heparin sodium produced by laboratory Hipolabor compared to heparin manufactured by APP in patients on hemodialysis due to renal failure, through the control of hemostasis, verified by formation of clot (fibrin) in the hemodialysis system and pharmacodynamic parameters (TTPA and Anti-Xa) during the use of heparin

ELIGIBILITY:
Inclusion Criteria:

1. Research that patients agreed to participate and signed the written informed consent;
2. Patients aged over 18 years, both sexes, regardless of color or social class;
3. Patients with impaired renal function in chronic hemodialysis schedule of at least 3 times a week and giving the use of heparin in the prophylaxis of thrombosis in the system.

Exclusion Criteria:

1. Hypersensitivity to heparin sodium and / or benzyl alcohol;
2. History of bleeding or disease that the change of blood coagulation could aggravate or terminate the clinical manifestations, such as tables of active peptic or gastric ulcer;
3. Severe liver disease;
4. Cancer;
5. Period of gestation;
6. Genetic abnormality of the coagulation system;
7. Multiple trauma;
8. Use of aspirin in high doses (above 200mg per day);
9. Use of glucocorticoids for at least 1 month;
10. Use of other anticoagulants;
11. Submission of a big surgery done less than 15 days;
12. History of persistent hypertension at the end of dialysis than 150/100 mmHg;
13. Indicated doses of heparin 20% above or below 150UI/kg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of heparin in thrombi formation. | 12 consecutive sessions
  During 4 weeks (3 times/week)of treatment will be avaluete thrombi formation in the dialysis system and decrease in net volume of the capillary dialyzer (primming) under formation of fibrin.

SECONDARY OUTCOMES:
Alteration of the pharmacodynamic parameters. | 12 consecutive sessions.
  During 4 weeks (3 times/week)of treatment will be avaluate evoluation fo TTPA and ANTI-XA.
Evaluation of Anti-Xa | 12 consecutive sessions (4 weeks - 3times/week)

CONTACTS AND LOCATIONS:
Locations (1):
- Lal Clinica Pesquisa E Desenvolvimento Ltda, Valinhos, São Paulo, Brazil